CLINICAL TRIAL: NCT01443845
Title: Study to Evaluate the Effect of Roflumilast 500 μg on Exacerbation Rate in Subjects With Chronic Obstructive Pulmonary Disease (COPD) Treated With a Fixed-Dose Combination of Long-Acting Beta Agonist and Inhaled Corticosteroid (LABA/ICS)
Brief Title: Roflumilast in Chronic Obstructive Pulmonary Disease (COPD) Patients Treated With Fixed Dose Combinations of Long-acting β2-agonist (LABA) and Inhaled Corticosteroid (ICS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROF-MD-07
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: COPD; COPD Exacerbation; Lung Diseases; Respiratory Disorders; Pulmonary Disease; Chronic Obstructive Lung Diseases; Chronic Obstructive Airway Disease
Keywords: COPD; Exacerbations; Roflumilast; Daliresp
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiration Disorders | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Roflumilast
  Interventions: Drug: Roflumilast
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Roflumilast 500 µg, oral administration, once per day
  Other Names: Daliresp
  Arms: 1
Drug: Placebo — Dose-matched placebo, oral administration, once per day.
  Arms: 2

SUMMARY:
To demonstrate the additional benefit of roflumilast when added on to fixed-dose combination (FDC) LABA/ICS in the reduction of exacerbations in subjects with severe to very severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients at least 40 years of age
* 2. History of COPD (according to Global Initiative for Chronic Obstructive Lung Disease [GOLD] 2010) for at least 12 months prior to Screening (Visit 1) associated with chronic productive cough for 3 months in each of 2 consecutive years (with other causes of productive cough excluded). Only patients with chronic bronchitis will be included (concomitant emphysema is permitted)
* 3. Forced expiratory volume after 1 second (FEV1)/forced vital capacity (FVC) ratio (postbronchodilator) < 70% at Screening (Visit 1)
* 4. FEV1 (postbronchodilator) ≤ 50% of predicted at Screening (Visit 1)
* 5. At least two documented moderate or severe COPD exacerbations within 12 months prior to Screening (Visit 1)
* 6. Patients must be on FDC LABA/ICS treatment ≥ 3 months prior to Screening (Visit 1)
* 7. Former smokers (defined as smoking cessation at least 1 year ago) or current smokers (including patients who ceased smoking within the past year) both with a smoking history of at least 20 pack-years

Exclusion Criteria:

* 1. Moderate or severe COPD exacerbation and/or COPD exacerbations treated with antibiotics or systemic glucocorticosteroids within 4 weeks of Screening (Visit 1) (ie, patients must be clinically stable)
* 2. Known alpha-1-antitrypsin deficiency
* 3. Current diagnosis of asthma (either controlled or uncontrolled) (Note: History of childhood asthma is not exclusionary.)
* 4. Body mass index (BMI) ≥ 45 kg/m2
* 5. Patients with a history (within 5 years) or current diagnosis of cancer other than basal or squamous cell skin cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2354 (Actual)
Dates: Start 2011-09-30 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (338):
- United States (217):
  - Forest Investigative Site 081, Anniston, Alabama
  - Forest Investigative Site 065, Athens, Alabama
  - Forest Investigative Site 131, Florence, Alabama
  - Forest Investigative Site 073, Mobile, Alabama
  - Forest Investigative Site 272, Mesa, Arizona
  - Forest Investigative Site 091, Peoria, Arizona
  - Forest Investigative Site 034, Phoenix, Arizona
  - Forest Investigative Site 188, Phoenix, Arizona
  - Forest Investigative Site 211, Phoenix, Arizona
  - Forest Investigative Site 247, Phoenix, Arizona
  - Forest Investigative Site 208, Fort Smith, Arkansas
  - Forest Investigative Site 101, Little Rock, Arkansas
  - Forest Investigative Site 074, Bellflower, California
  - Forest Investigative Site 060, Fresno, California
  - Forest Investigative Site 329, Fresno, California
  - Forest Investigative Site 245, Fullerton, California
  - Forest Investigative Site 310, Garden Grove, California
  - Forest Investigative Site 297, Lakewood, California
  - Forest Investigative Site 116, Long Beach, California
  - Forest Investigative Site 085, Los Angeles, California
  - Forest Investigative Site 241, Los Angeles, California
  - Forest Investigative Site 299, Northridge, California
  - Forest Investigative Site 213, Palo Alto, California
  - Forest Investigative Site 268, Pismo Beach, California
  - Forest Investigative Site 025, Riverside, California
  - Forest Investigative Site 143, Roseville, California
  - Forest Investigative Site 104, Sacramento, California
  - Forest Investigative Site 352, San Diego, California
  - Forest Investigative Site 038, San Diego, California
  - Forest Investigative Site 326, San Jose, California
  - Forest Investigative Site 209, Torrance, California
  - Forest Investigative Site 331, Stamford, Connecticut
  - Forest Investigative Site 017, Waterbury, Connecticut
  - Forest Investigative Site 124, Newark, Delaware
  - Forest Investigative Site 196, Brandon, Florida
  - Forest Investigative Site 224, Brandon, Florida
  - Forest Investigative Site 358, Brandon, Florida
  - Forest Investigative Site 166, Chiefland, Florida
  - Forest Investigative Site 111, Clearwater, Florida
  - Forest Investigative Site 123, Clearwater, Florida
  - Forest Investigative Site 291, Coral Gables, Florida
  - Forest Investigative Site 239, DeFuniak Springs, Florida
  - Forest Investigative Site 001, Fort Lauderdale, Florida
  - Forest Investigative Site 165, Fort Walton Beach, Florida
  - Forest Investigative Site 102, Gainesville, Florida
  - Forest Investigative Site 003, Hollywood, Florida
  - Forest Investigative Site 023, Jacksonville, Florida
  - Forest Investigative Site 077, Kissimmee, Florida
  - Forest Investigative Site 330, Kissimmee, Florida
  - Forest Investigative Site 027, Miami, Florida
  - Forest Investigative Site 229, Miami, Florida
  - Forest Investigative Site 115, Miami, Florida
  - Forest Investigative Site 339, Miami, Florida
  - Forest Investigative Site 092, Naples, Florida
  - Forest Investigative Site 004, Orlando, Florida
  - Forest Investigative Site 187, Ormond Beach, Florida
  - Forest Investigative Site 069, Pensacola, Florida
  - Forest Investigative Site 161, Ponte Vedra, Florida
  - Forest Investigative Site 087, Port Orange, Florida
  - Forest Investigative Site 109, Saint Cloud, Florida
  - Forest Investigative Site 121, St. Petersburg, Florida
  - Forest Investigative Site 357, St. Petersburg, Florida
  - Forest Investigative Site 002, Tamarac, Florida
  - Forest Investigative Site 287, Tampa, Florida
  - Forest Investigative Site 052, Tampa, Florida
  - Forest Investigative Site 011, Winter Park, Florida
  - Forest Investigative Site 348, Winter Park, Florida
  - Forest Investigative Site 103, Canton, Georgia
  - Forest Investigative Site 292, Dawsonville, Georgia
  - Forest Investigative Site 042, Duluth, Georgia
  - Forest Investigative Site 140, Gainesville, Georgia
  - Forest Investigative Site 030, Lawrenceville, Georgia
  - Forest Investigative Site 321, Woodstock, Georgia
  - Forest Investigative Site 008, Coeur d'Alene, Idaho
  - Forest Investigative Site 119, Eagle, Idaho
  - Forest Investigative Site 201, Bolingbrook, Illinois
  - Forest Investigative Site 206, Downers Grove, Illinois
  - Forest Investigative Site 136, Elk Grove Village, Illinois
  - Forest Investigative Site 139, Oak Lawn, Illinois
  - Forest Investigative Site 227, Peoria, Illinois
  - Forest Investigative Site 334, Springfield, Illinois
  - Forest Investigative Site 263, Elwood, Indiana
  - Forest Investigative Site 342, Lafayette, Indiana
  - Forest Investigative Site 293, Michigan City, Indiana
  - Forest Investigative Site 264, Muncie, Indiana
  - Forest Investigative Site 135, Council Bluffs, Iowa
  - Forest Investigative Site 256, Iowa City, Iowa
  - Forest Investigative Site 214, Olathe, Kansas
  - Forest Investigative Site 316, Topeka, Kansas
  - Forest Investigative Site 301, Wichita, Kansas
  - Forest Investigative Site 051, Bowling Green, Kentucky
  - Forest Investigative Site 075, Crescent Springs, Kentucky
  - Forest Investigative Site 351, Hazard, Kentucky
  - Forest Investigative Site 068, Lexington, Kentucky
  - Forest Investigative Site 088, Louisville, Kentucky
  - Forest Investigative Site 053, Owensboro, Kentucky
  - Forest Investigative Site 273, Lafayette, Louisiana
  - Forest Investigative Site 070, Opelousas, Louisiana
  - Forest Investigative Site 097, Sunset, Louisiana
  - Forest Investigative Site 128, Lewiston, Maine
  - Forest Investigative Site 248, Baltimore, Maryland
  - Forest Investigative Site 020, Columbia, Maryland
  - Forest Investigative Site 072, Towson, Maryland
  - Forest Investigative Site 106, Fall River, Massachusetts
  - Forest Investigative Site 044, North Dartmouth, Massachusetts
  - Forest Investigative Site 350, Pittsfield, Massachusetts
  - Forest Investigative Site 157, Ann Arbor, Michigan
  - Forest Investigative Site 341, Detroit, Michigan
  - Forest Investigative Site 328, Kalamazoo, Michigan
  - Forest Investigative Site 063, Livonia, Michigan
  - Forest Investigative Site 322, Saint Joseph, Michigan
  - Forest Investigative Site 303, Edina, Minnesota
  - Forest Investigative Site 056, Fridley, Minnesota
  - Forest Investigative Site 082, Rochester, Minnesota
  - Forest Investigative Site 033, Chesterfield, Missouri
  - Forest Investigative Site 098, Saint Charles, Missouri
  - Forest Investigative Site 117, Springfield, Missouri
  - Forest Investigative Site 186, St Louis, Missouri
  - Forest Investigative Site 288, St Louis, Missouri
  - Forest Investigative Site 333, Butte, Montana
  - Forest Investigative Site 029, Missoula, Montana
  - Forest Investigative Site 197, Bellevue, Nebraska
  - Forest Investigative Site 267, Fremont, Nebraska
  - Forest Investigative Site 337, Fremont, Nebraska
  - Forest Investigative Site 315, Lincoln, Nebraska
  - Forest Investigative Site 108, Lincoln, Nebraska
  - Forest Investigative Site 345, Omaha, Nebraska
  - Forest Investigative Site 079, Henderson, Nevada
  - Forest Investigative Site 270, Henderson, Nevada
  - Forest Investigative Site 067, Cherry Hill, New Jersey
  - Forest Investigative Site 327, Clifton, New Jersey
  - Forest Investigative Site 144, Hackensack, New Jersey
  - Forest Investigative Site 317, Summit, New Jersey
  - Forest Investigative Site 226, Brooklyn, New York
  - Forest Investigative Site 199, Great Neck, New York
  - Forest Investigative Site 071, New York, New York
  - Forest Investigative Site 013, Rochester, New York
  - Forest Investigative Site 066, Syracuse, New York
  - Forest Investigative Site 158, West Seneca, New York
  - Forest Investigative Site 313, Asheville, North Carolina
  - Forest Investigative Site 193, Burlington, North Carolina
  - Forest Investigative Site 142, Charlotte, North Carolina
  - Forest Investigative Site 259, Charlotte, North Carolina
  - Forest Investigative Site 019, Elizabeth City, North Carolina
  - Forest Investigative Site 318, Shelby, North Carolina
  - Forest Investigative Site 078, Shelby, North Carolina
  - Forest Investigative Site 176, Wilmington, North Carolina
  - Forest Investigative Site 282, Winston-Salem, North Carolina
  - Forest Investigative Site 314, Winston-Salem, North Carolina
  - Forest Investigative Site 164, Canton, Ohio
  - Forest Investigative Site 149, Cincinnati, Ohio
  - Forest Investigative Site 061, Cincinnati, Ohio
  - Forest Investigative Site 040, Cincinnati, Ohio
  - Forest Investigative Site 280, Cincinnati, Ohio
  - Forest Investigative Site 009, Columbus, Ohio
  - Forest Investigative Site 353, Dayton, Ohio
  - Forest Investigative Site 059, Marion, Ohio
  - Forest Investigative Site 154, Marion, Ohio
  - Forest Investigative Site 346, Toledo, Ohio
  - Forest Investigative Site 105, Zanesville, Ohio
  - Forest Investigative Site 167, Oklahoma City, Oklahoma
  - Forest Investigative Site 281, Oklahoma City, Oklahoma
  - Forest Investigative Site 236, Tulsa, Oklahoma
  - Forest Investigative Site 285, Medford, Oregon
  - Forest Investigative Site 289, Portland, Oregon
  - Forest Investigative Site 218, Portland, Oregon
  - Forest Investigative Site 086, Altoona, Pennsylvania
  - Forest Investigative Site 340, Beaver, Pennsylvania
  - Forest Investigative Site 120, Downingtown, Pennsylvania
  - Forest Investigative Site 062, Erie, Pennsylvania
  - Forest Investigative Site 277, Norristown, Pennsylvania
  - Forest Investigative Site 230, Philadelphia, Pennsylvania
  - Forest Investigative Site 205, Philadelphia, Pennsylvania
  - Forest Investigative Site 336, Pittsburgh, Pennsylvania
  - Forest Investigative Site 364, Pittsburgh, Pennsylvania
  - Forest Investigative Site 344, Pittsburgh, Pennsylvania
  - Forest Investigative Site 010, Tipton, Pennsylvania
  - Forest Investigative Site 064, Uniontown, Pennsylvania
  - Forest Investigative Site 228, Johnston, Rhode Island
  - Forest Investigative Site 283, Lincoln, Rhode Island
  - Forest Investigative Site 365, Providence, Rhode Island
  - Forest Investigative Site 305, Charleston, South Carolina
  - Forest Investigative Site 093, Easley, South Carolina
  - Forest Investigative Site 257, Fort Mill, South Carolina
  - Forest Investigative Site 233, Gaffney, South Carolina
  - Forest Investigative Site 110, Greenville, South Carolina
  - Forest Investigative Site 300, Pelzer, South Carolina
  - Forest Investigative Site 204, Rock Hill, South Carolina
  - Forest Investigative Site 021, Spartanburg, South Carolina
  - Forest Investigative Site 012, Union, South Carolina
  - Forest Investigative Site 058, Rapid City, South Dakota
  - Forest Investigative Site 223, Bristol, Tennessee
  - Forest Investigative Site 050, Fayetteville, Tennessee
  - Forest Investigative Site 253, Shelbyville, Tennessee
  - Forest Investigative Site 024, Arlington, Texas
  - Forest Investigative Site 177, Boerne, Texas
  - Forest Investigative Site 090, Corsicana, Texas
  - Forest Investigative Site 172, Dallas, Texas
  - Forest Investigative Site 237, Houston, Texas
  - Forest Investigative Site 271, Houston, Texas
  - Forest Investigative Site 370, Houston, Texas
  - Forest Investigative Site 195, Houston, Texas
  - Forest Investigative Site 312, Houston, Texas
  - Forest Investigative Site 332, Huntsville, Texas
  - Forest Investigative Site 232, Longview, Texas
  - Forest Investigative Site 049, Tyler, Texas
  - Forest Investigative Site 181, Colchester, Vermont
  - Forest Investigative Site 125, Abingdon, Virginia
  - Forest Investigative Site 202, Richmond, Virginia
  - Forest Investigative Site 231, Richmond, Virginia
  - Forest Investigative Site 045, Richmond, Virginia
  - Forest Investigative Site 184, Spokane, Washington
  - Forest Investigative Site 174, Spokane, Washington
  - Forest Investigative Site 217, Tacoma, Washington
  - Forest Investigative Site 335, Charleston, West Virginia
  - Forest Investigative Site 319, Morgantown, West Virginia
  - Forest Investigative Site 146, West Allis, Wisconsin
- Argentina (20):
  - Forest Investigative Site 403, Buenos Aires, Buenos Aires
  - Forest Investigative Site 418, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Forest Investigative Site 402, Florida, Buenos Aires
  - Forest Investigative Site 405, La Plata, Buenos Aires
  - Forest Investigative Site 406, Lanús Este, Buenos Aires
  - Forest Investigative Site 413, Mar del Plata, Buenos Aires
  - Forest Investigative Site 407, Paraná, Entre Ríos Province
  - Forest Investigative Site 404, Mendoza, Mendoza Province
  - Forest Investigative Site 412, Rosario, Santa Fe Province
  - Forest Investigative Site 409, Rosario, Santa Fe Province
  - Forest Investigative Site 411, Buenos Aires
  - Forest Investigative Site 414, Buenos Aires
  - Forest Investigative Site 419, Buenos Aires
  - Forest Investigative Site 416, Buenos Aires
  - Forest Investigative Site 415, Derqui Pilar - Buenos Aires
  - Forest Investigative Site 417, La Plata
  - Forest Investigative Site 420, Mendoza
  - Forest Investigative Site 410, San Juan Bautista
  - Forest Investigative Site 401, San Miguel de Tucumán
  - Forest Investigative Site 408, Santa Fe
- Canada (5):
  - Forest Investigative Site 235, Calgary, Alberta
  - Forest Investigative Site 162, North Vancouver, British Columbia
  - Forest Investigative Site 302, Burlington, Ontario
  - Forest Investigative Site 185, Montreal, Quebec
  - Forest Investigative Site 127, Saskatoon, Saskatchewan
- Forest Investigative Site 421, Talcahuano, Chile
- Colombia (2):
  - Forest Investigative Site 442, Bogotá
  - Forest Investigative Site 443, Bogotá
- Italy (2):
  - Forest Investigative Site 461, Chieti
  - Forest Investigative Site 464, Roma
- Malaysia (4):
  - Forest Investigative Site 505, Batu Caves
  - Forest Investigative Site 501, Kuala Lumpur
  - Forest Investigative Site 504, Kuala Lumpur
  - Forest Investigative Site 502, Kuantan
- Mexico (4):
  - Forest Investigative Site 522, Monterrey, Nuevo León
  - Forest Investigative Site 526, Mérida, Yucatán
  - Forest Investigative Site 524, Guadalajara
  - Forest Investigative Site 521, Monterrey
- Peru (8):
  - Forest Investigative Site 543, Bellavista
  - Forest Investigative Site 550, Lima
  - Forest Investigative Site 551, Lima
  - Forest Investigative Site 545, Lima
  - Forest Investigative Site 546, Lima
  - Forest Investigative Site 549, Lima
  - Forest Investigative Site 544, Lima
  - Forest Investigative Site 541, Pueblo Libre
- Philippines (9):
  - Forest Investigative Site 569, Cavite
  - Forest Investigative Site 567, Iloilo City
  - Forest Investigative Site 568, Iloilo City
  - Forest Investigative Site 565, Manila
  - Forest Investigative Site 563, Pasig
  - Forest Investigative Site 562, Quezon City
  - Forest Investigative Site 564, Quezon City
  - Forest Investigative Site 566, Quezon City
  - Forest Investigative Site 561, Quezon City
- Romania (8):
  - Forest Investigative Site 585, Brasov
  - Forest Investigative Site 586, Bucharest
  - Forest Investigative Site 587, Bucharest
  - Forest Investigative Site 588, Bucharest
  - Forest Investigative Site 584, Bucharest
  - Forest Investigative Site 582, Bucharest
  - Forest Investigative Site 581, Iași
  - Forest Investigative Site 583, Iași
- Russia (17):
  - Forest Investigative Site 608, Barnaul
  - Forest Investigative Site 602, Kazan'
  - Forest Investigative Site 618, Kemerovo
  - Forest Investigative Site 609, Krasnodar
  - Forest Investigative Site 614, Krasnoyarsk
  - Forest Investigative Site 617, Moscow
  - Forest Investigative Site 605, Novosibirsk
  - Forest Investigative Site 606, Saint Petersburg
  - Forest Investigative Site 612, Saint Petersburg
  - Forest Investigative Site 619, Saint Petersburg
  - Forest Investigative Site 604, Saint Petersburg
  - Forest Investigative Site 611, Saint Petersburg
  - Forest Investigative Site 610, Saint Petersburg
  - Forest Investigative Site 601, Saint Petersburg
  - Forest Investigative Site 600, Saint Petersburg
  - Forest Investigative Site 607, Tomsk
  - Forest Investigative Site 620, Yaroslavl
- Serbia (7):
  - Forest Investigative Site 629, Knez-Selo, Nišava District
  - Forest Investigative Site 622, Belgrade
  - Forest Investigative Site 623, Belgrade
  - Forest Investigative Site 624, Belgrade
  - Forest Investigative Site 625, Belgrade
  - Forest Investigative Site 627, Kamenitz
  - Forest Investigative Site 628, Kragujevac
- Spain (3):
  - Forest Investigative Site 641, Cadiz
  - Forest Investigative Site 647, Loja
  - Forest Investigative Site 644, Salt
- Taiwan (4):
  - Forest Investigative Site 723, Kaohsiung Hsien
  - Forest Investigative Site 724, Puzih City
  - Forest Investigative Site 725, Taipei
  - Forest Investigative Site 722, Taipei
- Thailand (4):
  - Forest Investigative Site 662, Hat Yai, Changwat Songkhla
  - Forest Investigative Site 664, Bangkok
  - Forest Investigative Site 663, Bangkok
  - Forest Investigative Site 661, Muang
- Ukraine (23):
  - Forest Investigative Site 699, Cherkasy
  - Forest Investigative Site 691, Dnipropetrovsk
  - Forest Investigative Site 692, Donetsk
  - Forest Investigative Site 689, Donetsk
  - Forest Investigative Site 690, Ivano-Frankivsk
  - Forest Investigative Site 697, Kharkiv
  - Forest Investigative Site 693, Kharkiv
  - Forest Investigative Site 682, Kharkiv
  - Forest Investigative Site 709, Kremenchuk
  - Forest Investigative Site 698, Kyiv
  - Forest Investigative Site 683, Kyiv
  - Forest Investigative Site 684, Kyiv
  - Forest Investigative Site 687, Kyiv
  - Forest Investigative Site 685, Kyiv
  - Forest Investigative Site 681, Lviv
  - Forest Investigative Site 708, Mykolayiv
  - Forest Investigative Site 706, Poltava
  - Forest Investigative Site 695, Sumy
  - Forest Investigative Site 707, Vinnitsa
  - Forest Investigative Site 688, Zaporizhzhia
  - Forest Investigative Site 696, Zaporizhzhya
  - Forest Investigative Site 694, Zaporizhzhya
  - Forest Investigative Site 705, Zaporizhzhya

REFERENCES:
- [Derived] Martinez FJ, Rabe KF, Calverley PMA, Fabbri LM, Sethi S, Pizzichini E, McIvor A, Anzueto A, Alagappan VKT, Siddiqui S, Reisner C, Zetterstrand S, Roman J, Purkayastha D, Bagul N, Rennard SI. Determinants of Response to Roflumilast in Severe Chronic Obstructive Pulmonary Disease. Pooled Analysis of Two Randomized Trials. Am J Respir Crit Care Med. 2018 Nov 15;198(10):1268-1278. doi: 10.1164/rccm.201712-2493OC. PMID 29763572
- [Derived] Karpefors M, Weatherall J. The Tendril Plot-a novel visual summary of the incidence, significance and temporal aspects of adverse events in clinical trials. J Am Med Inform Assoc. 2018 Aug 1;25(8):1069-1073. doi: 10.1093/jamia/ocy016. PMID 29579254
- [Derived] Martinez FJ, Rabe KF, Sethi S, Pizzichini E, McIvor A, Anzueto A, Alagappan VK, Siddiqui S, Rekeda L, Miller CJ, Zetterstrand S, Reisner C, Rennard SI. Effect of Roflumilast and Inhaled Corticosteroid/Long-Acting beta2-Agonist on Chronic Obstructive Pulmonary Disease Exacerbations (RE(2)SPOND). A Randomized Clinical Trial. Am J Respir Crit Care Med. 2016 Sep 1;194(5):559-67. doi: 10.1164/rccm.201607-1349OC. PMID 27585384
- See also: RESPOND Protocol_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14667&filename=RESPOND%20Protocol_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from September 2011 to October 2014 for a total of 380 study centers screened patients for the study: Italy, Spain, United States, Ukraine, Argentina, Russia, Philippines, Romania, Serbia, Canada, Malaysia, Thailand, Mexico, Peru and Taiwan.
Pre-assignment Details: The study consisted of 2 weeks of single-blind placebo lead-in with fixed-dose combination (FDC) long-acting β2-agonist(s) (LABA)/inhaled corticosteroid(s) (ICS) treatment followed by 52 weeks of double-blind treatment in addition to maintenance FDC LABA/ICS.
Period: Overall Study
Arm/Group | Placebo | Roflumilast
Started | 1176 | 1178
Completed | 922 | 841
Not Completed | 254 | 337
Not completed — Protocol Violation | 43 | 45
Not completed — Other reasons, such as COPD exacerbation | 44 | 44
Not completed — Deterioration in pulmonary function | 1 | 4
Not completed — Lack of Efficacy | 10 | 5
Not completed — Adverse Event | 64 | 138
Not completed — Withdrawal by Subject | 63 | 67
Not completed — Military Conflict - Site Terminated | 20 | 21
Not completed — Lost to Follow-up | 9 | 13

BASELINE CHARACTERISTICS:
Population: The demographic information provided here is for the safety population. The safety population (numbering 2352 patients) of the trial does not include 2 patients from the enrolled population (numbering 2354 patients), due to a protocol deviation for one patient and an adverse event for a second patient, both in the placebo arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Roflumilast | Total
Number analyzed (Participants) | 1174 | 1178 | 2352
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.4) | 64.4 (8.8) | 64.5 (8.6)
Age, Customized [Number; unit: Participants]
  Adults 40-65 years | 634 | 640 | 1274
  Adults over 65 years | 540 | 538 | 1078
Sex/Gender, Customized [Number; unit: Participants]
  Male | 794 | 821 | 1615
  Female | 380 | 357 | 737
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 944 | 935 | 1879
  Black or African American | 27 | 35 | 62
  Asian | 170 | 167 | 337
  American Indian or Alaska Native | 6 | 16 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Other | 27 | 23 | 50
Region of Enrollment [Number; unit: participants]
  Colombia | 7 | 10 | 17
  Argentina | 197 | 198 | 395
  Russian Federation | 77 | 77 | 154
  Romania | 55 | 54 | 109
  United States | 458 | 457 | 915
  Philippines | 130 | 131 | 261
  Ukraine | 95 | 95 | 190
  Malaysia | 6 | 7 | 13
  Thailand | 18 | 16 | 34
  Spain | 6 | 6 | 12
  Canada | 14 | 15 | 29
  Taiwan | 7 | 6 | 13
  Italy | 0 | 1 | 1
  Mexico | 22 | 22 | 44
  Serbia | 47 | 47 | 94
  Peru | 35 | 36 | 71
Ethnicity [Number; unit: Participants]
  Hispanic or Latino | 272 | 268 | 540
  Not Hispanic or Latino | 902 | 910 | 1812
ICS/LABA Therapy [Number; unit: Participants]
  Advair | 766 | 768 | 1534
  Symbicort | 408 | 410 | 818
Long-acting muscarinic antagonist(s) (LAMA) use [Number; unit: Participants]
  LAMA | 546 | 548 | 1094
  No-LAMA | 628 | 630 | 1258
BMI Category [Number; unit: Participants]
  Under weight: < 18.5 | 95 | 100 | 195
  Normal weight: >= 18.5 to < 25 | 480 | 468 | 948
  Over weight: >= 25 to < 30 | 347 | 342 | 689
  Obese: >= 30 | 252 | 268 | 520
Weight [Mean (Standard Deviation); unit: kg] | 72.57 (18.67) | 73.63 (19.57) | 73.10 (19.13)
Height [Median (Standard Deviation); unit: cm] | 167.53 (9.39) | 167.80 (9.35) | 167.67 (9.37)
Body-Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 25.72 (5.72) | 25.99 (5.91) | 25.86 (5.82)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate or Severe COPD Exacerbations Per Patient Per Year.
Description: Rate of moderate or severe COPD exacerbations, defined as requiring oral or parenteral glucocorticosteroids (moderate) or requiring hospitalization and/or leading to death (severe), during the double-blind treatment period.
Time Frame: Baseline to Week 52
Population: Intent-to-Treat Study Population
Measure: Number (95% Confidence Interval); unit: COPD exacerbations per patient per year
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 1174 | 1178
COPD exacerbations per patient per year | 1.27 [1.17 to 1.39] | 1.17 [1.06 to 1.28]
Statistical Analysis 1: Comparison: Placebo vs Roflumilast; Rate ratio (Roflumilast/Placebo). A rate ratio < 1 represents a favorable outcome for the test treatment; Test type: Superiority or Other; p = 0.1634, negative binomial regression; Rate Ratio = 0.92, 95% CI 2-sided [0.81 to 1.04], Standard Error of Mean 0.063 — p-values are based on a negative binomial regression with factors Treatment and LAMA use
Statistical Analysis 2: Comparison: Placebo vs Roflumilast; Subgroup Analysis - By Sex - Male; Test type: Superiority or Other; p = 0.0195, negative binomial regression; Rate Ratio = 0.83, 95% CI 2-sided [0.71 to 0.97], Standard Error of Mean 0.08
Statistical Analysis 3: Comparison: Placebo vs Roflumilast; Subgroup Analysis - By Sex - Female; Test type: Superiority or Other; p = 0.3164, negative binomial regression; Rate Ratio = 1.11, 95% CI 2-sided [0.91 to 1.35], Standard Error of Mean 0.101
Statistical Analysis 4: Comparison: Placebo vs Roflumilast; Subgroup analysis between patients taking Advair verses patients taking Symbicort as LABA/ICS therapy; Test type: Superiority or Other; p = 0.0385, negative binomial regression; Rate Ratio = 0.85, 95% CI 2-sided [0.74 to 0.99], Standard Error of Mean 0.076
Statistical Analysis 5: Comparison: Placebo vs Roflumilast; Subgroup analysis between patients taking Advair verses patients taking Symbicort as LABA/ICS therapy; Test type: Superiority or Other; p = 0.6475, negative binomial regression; Rate Ratio = 1.05, 95% CI 2-sided [0.84 to 1.32], Standard Error of Mean 0.114

2. Secondary Outcome: Rate of COPD Exacerbations That Led to Hospitalization or Death (ie, Severe COPD Exacerbations)
Description: Rate of moderate or severe COPD exacerbations, defined as requiring hospitalization and/or leading to death (severe), during the double-blind treatment period.
Time Frame: Week 0 (Visit 2) to Week 52
Population: Intent-to-Treat Study Population
Measure: Number (95% Confidence Interval); unit: COPD exacerbations per patient per year
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 1174 | 1178
COPD exacerbations per patient per year | 0.29 [0.25 to 0.34] | 0.28 [0.23 to 0.33]
Statistical Analysis 1: Comparison: Placebo vs Roflumilast; Test type: Superiority or Other; p = 0.6354, negative binomial regression; Rate Ratio = 0.95, 95% CI 2-sided [0.75 to 1.19], Standard Error of Mean 0.118

3. Secondary Outcome: Rate of Moderate or Severe COPD Exacerbations or COPD Exacerbations Treated With Antibiotics
Description: Rate of moderate or severe COPD exacerbations treated with antibiotics during the double-blind treatment period.
Time Frame: Week 0 (Visit 2) to Week 52
Measure: Number (95% Confidence Interval); unit: COPD Exacerbations per Patient per Year
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 1174 | 1178
COPD Exacerbations per Patient per Year | 1.45 [1.34 to 1.57] | 1.31 [1.20 to 1.43]
Statistical Analysis 1: Comparison: Placebo vs Roflumilast; Test type: Superiority or Other; p = 0.0884, negative binomial regression; Rate Ratio = 0.9, 95% CI 2-sided [0.8 to 1.02], Standard Error of Mean 0.06

4. Secondary Outcome: Mean Change in Predose Forced Expiratory Volume in 1 Second (FEV1)
Description: Mean change from randomization (Visit 2) over 52 weeks of treatment in predose forced expiratory volume in 1 second (FEV1)
Time Frame: Week 0 (Visit 2) to Week 52
Population: Intent-to-Treat Population who the completed 52-week treatment period
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | Roflumilast
Number analyzed (Participants) | 1105 | 1054
Liters | -0.0091 (0.0047) | 0.0441 (0.0048)
Statistical Analysis 1: Comparison: Placebo vs Roflumilast; Test type: Superiority or Other; p < 0.0001, Mixed Model for Repeated Measures (MMRM) — The MMRM analysis is based on all postbaseline observed data using a mixed model with terms for treatment, baseline, visit, LAMA use, treatment-by-visit and baseline-by-visit interactions; Mean Difference (Final Values) = 0.0532, 95% CI 2-sided [0.04 to 0.0664], Standard Error of Mean 0.0067

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the start of the 52-week double-blind treatment period, to 30 days after the end of treatment.
Arm/Group | Placebo | Roflumilast
Serious Adverse Events (participants affected / at risk) | 162/1174 | 180/1178
Other Adverse Events (participants affected / at risk) | 188/1174 | 317/1178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=1174) | Roflumilast (N=1178)
Aortic aneurysm (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 2 | 3
Angiodysplasia (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 0
Intra-abdominal haematoma (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenosquamous cell lung cancern (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer limited stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/380 | 0/357
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/794 | 0/821
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/380 | 0/357
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 6
Incarcerated hernia (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Death (General disorders) | 3 | 0
Fatigue (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Adnexa uteri mass (Reproductive system and breast disorders) | 1/380 | 0/357
Adnexal torsion (Reproductive system and breast disorders) | 1/380 | 0/357
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/794 | 0/821
Fall (Injury, poisoning and procedural complications) | 4 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Tinea pedis (Investigations) | 1 | 0
Nutritional condition abnormal (Investigations) | 0 | 1
Weight increased (Investigations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 7
Cardiac arrest (Cardiac disorders) | 0 | 5
Atrial fibrillation (Cardiac disorders) | 5 | 4
Angina pectoris (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 3 | 3
Cardiogenic shock (Cardiac disorders) | 0 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 3
Angina unstable (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 3 | 2
Myocardial infarction (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 2 | 1
Cor pulmonale acute (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Myocardial rupture (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Choledochal cyst (Congenital, familial and genetic disorders) | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Cervical radiculopathy (Nervous system disorders) | 0/380 | 1/357
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 3
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Hyphaema (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Mydriasis (Eye disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 0 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonia (Infections and infestations) | 45 | 47
Sepsis (Infections and infestations) | 4 | 3
Gastroenteritis (Infections and infestations) | 1 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 2
Amoebic dysentery (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 7 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Chronic hepatitis C (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tracheobronchitis viral (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1174) | Roflumilast (N=1178)
Weight decreased (Investigations) | 27 | 91
Headache (Nervous system disorders) | 48 | 80
Diarrhoea (Gastrointestinal disorders) | 36 | 119
Nausea (Gastrointestinal disorders) | 30 | 62
Upper respiratory tract infection (Infections and infestations) | 66 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other